CLINICAL TRIAL: NCT01807572
Title: Relation of Consummatory and Anticipatory Food Reward to Obesity
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK080760-01
Record Dates: First submitted 2013-02-07; First posted 2013-03-08 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Weight Gain; Food Habits
MeSH Terms: conditions — Weight Gain; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All DNA samples will be stored at the Sequencing and Genomics lab of the University of Colorado. Only authorized staff will have access to remove the DNA samples for analysis. The DNA samples will be analyzed in this lab using standard DNA procedures. Data will be kept on the password protected server for a period of six months. After six months, the data will be destroyed. The DNA samples will be stored with a unique identification number, connected to a code list accessed only by our research team. Once the analysis has been completed, the saliva sample will be destroyed by soaking it in bleach. This will remove all DNA. In addition, by the end of the study the code list connecting subject numbers with DNA numbers will be destroyed. No individual samples, analyzed results, or any other individual data will be shared with other researchers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- obesity risk status: Lean adolescents at high-risk for obesity, by virtue of parental obesity, and lean adolescents at low-risk for obesity, by virtue of lean parents.

SUMMARY:
Obesity is associated with increased risk for mortality, atherosclerotic cerebrovascular disease, coronary heart disease, colorectal cancer, hyperlipidemia, hypertension, gallbladder disease, and diabetes mellitus, resulting in over 111,000 deaths annually in the United States ). In the US, 65% of adults are overweight or obese. Unfortunately, the treatment of choice for obesity (behavioral weight loss treatment) only results in a 10% reduction in body weight on average and most patients regain this weight within a few years. Further, most obesity prevention programs do not reduce risk for future weight gain. The limited success of treatment and prevention interventions may be due to an incomplete understanding of the processes that increase risk for obesity. Recent data suggest that obese adults show abnormalities in reward from food intake and anticipated food intake relative to lean adults, but the precise nature of these abnormalities is unclear and it has not been established whether these abnormalities predate obesity onset or are a consequence. It is vital to elucidate risk factors for obesity onset to advance understanding of etiological processes and determine the content of prevention and treatment programs.

The goals of this study are to (1) determine whether adolescents at high-risk for obesity, by virtue of having two obese parents, show abnormalities in reward from food intake (consummatory food reward) and anticipated reward from food intake (anticipatory food reward) compared to adolescents who are at low-risk for obesity, (2) determine whether abnormalities in consummatory and anticipatory food reward increase risk for weight gain and obesity onset, (3) examine moderators that may amplify the relations of consummatory and anticipatory food reward to unhealthy weight gain, and (4) examine changes in consummatory and anticipatory food reward in those participants who show obesity onset relative to those not showing obesity onset. Each of these goals is described in more detail below.

ELIGIBILITY:
Inclusion Criteria:

* We will require that adolescents have age- and sex- adjusted standardized body mass index (BMI) scores between the 25th and 75th percentile at baseline for inclusion.
* Low risk youth: Lean parents will have a BMI between 18 and 25.
* High risk youth: Obese parents will have a BMI value of greater than 30.

Exclusion Criteria:

* Students who report contraindicators of fMRI (e.g., metal implants, braces, or pregnancy).
* Current major psychiatric disorders (including substance use disorders, conduct disorder, oppositional defiant disorder, ADHD, major depression, bipolar disorder, panic disorder, agoraphobia, or generalized anxiety disorder)
* Current use of analgesics and other psychoactive drugs (e.g., cocaine)
* Serious medical complications (e.g., diabetes)
* Relevant food allergies
* Current smoking
* Current weight loss dieting

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be 140 lean adolescents at risk for obesity (by virtue of having two obese parents) and 40 lean adolescents with two lean parents. Participants will range in age from 14-16 and be recruited from high schools.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2009-06; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Test whether high-risk youth show abnormalities in consummatory and anticipatory food reward relative to low-risk youth | up to 3 years
  Using fMRI to test whether high-risk youth for obesity show differential neural responses in the striatum, and oral somatosensory and gustatory related brain regions when anticipating and during intake of a palatable food, relative to youth at low risk for obesity.

SECONDARY OUTCOMES:
Test the hypothesis that individuals showing abnormalities in anticipatory and consummatory food reward are at increased risk for future weight gain and obesity onset over a 3-year follow-up | up to 3 years
  Determine whether those showing hyper-brain activation during anticipation and intake of a palatable food (via fMRI) gain more body weight over a three year period.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Winter SR, Yokum S, Stice E, Osipowicz K, Lowe MR. Elevated reward response to receipt of palatable food predicts future weight variability in healthy-weight adolescents. Am J Clin Nutr. 2017 Apr;105(4):781-789. doi: 10.3945/ajcn.116.141143. Epub 2017 Feb 22. PMID 28228422
- [Derived] Burger KS, Stice E. Elevated energy intake is correlated with hyperresponsivity in attentional, gustatory, and reward brain regions while anticipating palatable food receipt. Am J Clin Nutr. 2013 Jun;97(6):1188-94. doi: 10.3945/ajcn.112.055285. Epub 2013 Apr 17. PMID 23595877